CLINICAL TRIAL: NCT05867329
Title: A Sequential Multiple Assignment Randomized Trial (SMART) Feasibility Pilot Developing and Optimizing Patient-Tailored Adaptive Treatment Strategies (ATS) for Acute Severe Ulcerative Colitis (ASUC)
Brief Title: Feasibility Pilot Sequential Multiple Assignment Randomized Trial (SMART) for Acute Severe Ulcerative Colitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Berinstein, Jeffrey (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Berinstein, Jeffrey, Assistant Professor Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HUM00228245; 1K23DK134764-01 (NIH)
Record Dates: First submitted 2023-04-18; First posted 2023-05-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Ulcerative Colitis Acute
Keywords: Acute Severe Ulcerative Colitis; Ulcerative colitis flare
MeSH Terms: interventions — Cyclosporine; upadacitinib; Methylprednisolone Hemisuccinate; Prednisone

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to stage 1 and then be evaluated day 3. If patients are non-responders (defined by protocol) re-randomization for the second stage will take place. Patients that are responders at day 3 will continue with stage 1 treatment. Response to the second-stage of treatment will be calculated 72 hours after initiation of second-stage treatment and on every day up to day 10. If a patient meets any of the second-stage treatment failure criteria (per protocol) on day 6 through day 10, the patient will be considered to have failed second-stage therapy and will be referred for colectomy. If a patient does not meet criteria for second-stage treatment failure or criteria for safe discharge (see the protocol) the patient will be permitted to continue second-stage treatment for a maximum of 7 days (day 10 of intervention). Physicians care for patients enrolled in our study will be interviewed to evaluate acceptability and feasibility.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Methylprednisolone (Experimental): Methylprednisolone Intravenous (IV) 30 milligram (mg) twice a day (BID)
  Interventions: Drug: Intravenous Methylprednisolone; Drug: Prednisone Oral Product
- Methylprednisolone plus Upadacitinib (Experimental): Methylprednisolone IV 30mg BID plus Upadacitinib 45mg every day.
  Interventions: Drug: Upadacitinib Extended Release Oral Tablet; Drug: Intravenous Methylprednisolone
- Oral Upadacitinib (Experimental): Upadacitinib 30 mg BID
  Interventions: Drug: Upadacitinib Extended Release Oral Tablet
- Methylprednisolone then Cyclosporine (Experimental): Methylprednisolone IV 30 mg BID Stage 1 and if determined to be a non-responder to Methylprednisolone, patient will receive rescue Cyclosporine (2milligram/kilogram (mg/kg) per day aiming for levels 200-400 nanograms per milliliter (ng/mL)) in addition to continuing Methylprednisolone for stage 2.
  Interventions: Drug: Cyclosporine Injection (IV); Drug: Cyclosporine Oral Product; Drug: Intravenous Methylprednisolone
- Methylprednisolone then Upadacitinib (Experimental): Methylprednisolone IV 30mg twice a day Stage 1 and if determined to be a non-responder to Methylprednisolone, patient will receive rescue Upadacitinib 30mg BID in addition to continuing Methylprednisolone for stage 2
  Interventions: Drug: Upadacitinib Extended Release Oral Tablet; Drug: Intravenous Methylprednisolone
- Oral Upadacitinib then Methylprednisolone (Experimental): Oral Upadacitinib 30mg BID for stage 1 then for patients that are non-responders, add rescue Methylprednisolone IV 30mg twice a day in addition to continuing Upadacitinib for stage 2.
  Interventions: Drug: Upadacitinib Extended Release Oral Tablet; Drug: Intravenous Methylprednisolone; Drug: Prednisone Oral Product
- Oral Upadacitinib then Methylprednisolone plus cyclosporine infusion (Experimental): Upadacitinib 30 mg BID for stage 1. If a patient is a non-responder to Upadacitinib 30 mg, then the study team will stop Upadacitinib and initiate Methylprednisolone IV 30mg twice a day plus Cyclosporine (2 milligram/kilogram (mg/kg) per day aiming for levels 200-400 nanograms per milliliter (ng/mL)) for stage 2.
  Interventions: Drug: Upadacitinib Extended Release Oral Tablet; Drug: Intravenous Methylprednisolone; Drug: Prednisone Oral Product
- Methylprednisolone plus Upadacitinib then cyclosporine (Experimental): Methylprednisolone IV 30mg BID and Oral Upadacitinib 45mg everyday stage 1 and then Cyclosporine 2 mg/kg per day aiming for levels 200-400ng/mL for stage 2.
  Interventions: Drug: Cyclosporine Injection (IV); Drug: Cyclosporine Oral Product; Drug: Intravenous Methylprednisolone
- Methylprednisolone plus Upadacitinib then increased Upadacitinib (Experimental): Methylprednisolone IV 30mg BID and Oral Upadacitinib 45mg everyday stage 1 and if determined to be a non-responder to Methylprednisolone and 45 mg Oral Upadacitinib, patient will receive rescue Upadacitinib 30mg BID in addition to continuing Methylprednisolone for stage 2.
  Interventions: Drug: Upadacitinib Extended Release Oral Tablet; Drug: Intravenous Methylprednisolone; Drug: Prednisone Oral Product

INTERVENTIONS:
Drug: Cyclosporine Injection (IV) — Drug be administered as weight-based continuous infusion (2mg/kg/day) during the second stage of treatment (if applicable).
  Cyclosporine monitoring will take place approximately 18-24 hours stage of treatment (Day 4 at the earliest). The goal is to achieve whole blood levels of 300 (range 200-400) ng/ml with adjustments according to the table in the protocol. The intravenous cyclosporine dosage is rarely raised above 4 mg/kg/day, in rare patients that are fast metabolizers.
  Other Names: Sandimmune
  Arms: Methylprednisolone plus Upadacitinib then cyclosporine; Methylprednisolone then Cyclosporine
Drug: Cyclosporine Oral Product — Once participants meet discharge criteria, participant's that received IV Cyclosporine (stage 2) will be transitioned to oral Cyclosporine.
  The oral dose is calculated to be approximately twice the daily intravenous dose or approximately 5 mg/kg, rounded to nearest 25 mg, and is administered every 12 hours (h). Oral cyclosporine solution will be administered as Sandimmune capsules available in 25mg 100mg capsules size.
  After the intervention period (during hospitalization after IV cyclosporine is complete) and during the follow-up period any cyclosporine adjustments are permissible under the current study protocol according to the discretion of the treating physician.
  Other Names: Sandimmune
  Arms: Methylprednisolone plus Upadacitinib then cyclosporine; Methylprednisolone then Cyclosporine
Drug: Upadacitinib Extended Release Oral Tablet — This will be administered orally once daily as 45mg (stage one) or twice daily as a 30mg oral tablet (first stage and second stage) of treatment (if applicable).
  Upon discharge a patient will be switched from Upadacitinib 30mg twice daily to 45mg daily for 8 weeks followed by 30mg or 15mg subsequently if Upadacitinib is to be continued after discharge. The choice of induction/maintenance agent initiated after discharge will be determined by inpatient treatment team and in consultation with the outpatient gastroenterologist. No patient will continue Upadacitinib 30mg twice daily after discharge from the hospital.
  Other Names: Rinvoq
  Arms: Methylprednisolone plus Upadacitinib; Methylprednisolone plus Upadacitinib then increased Upadacitinib; Methylprednisolone then Upadacitinib; Oral Upadacitinib; Oral Upadacitinib then Methylprednisolone; Oral Upadacitinib then Methylprednisolone plus cyclosporine infusion
Drug: Intravenous Methylprednisolone — Drug will be administered as 30mg twice daily during the first stage of treatment (if applicable) and through the second stage of treatment (if applicable). Prior to discharge a patient will be switched from IV Methylprednisolone to prednisone 40-60mg with plans to taper by 5mg/week (dose subject to adjustment by treating inpatient team and in consultation with the outpatient gastroenterologist).
  Other Names: Solu-Medrol
  Arms: Methylprednisolone; Methylprednisolone plus Upadacitinib; Methylprednisolone plus Upadacitinib then cyclosporine; Methylprednisolone plus Upadacitinib then increased Upadacitinib; Methylprednisolone then Cyclosporine; Methylprednisolone then Upadacitinib; Oral Upadacitinib then Methylprednisolone; Oral Upadacitinib then Methylprednisolone plus cyclosporine infusion
Drug: Prednisone Oral Product — Patients that received IV Methylprednisolone will be switched prior to discharge from IV Methylprednisolone to prednisone 40-60mg with plans to taper by 5mg/week (dose subject to adjustment by treating inpatient team and in consultation with the outpatient gastroenterologist).
  Other Names: Rayos
  Arms: Methylprednisolone; Methylprednisolone plus Upadacitinib then increased Upadacitinib; Oral Upadacitinib then Methylprednisolone; Oral Upadacitinib then Methylprednisolone plus cyclosporine infusion

SUMMARY:
The goal of this trial is to create personalized treatments for each patient admitted to the hospital with acute severe ulcerative colitis (ASUC). The study will test the feasibility and acceptability of these treatment strategies among patients and physicians so that the study team can later do a larger trial to test whether the medication treatment pathways help patients avoid colectomy while ensuring patient's are safe.

DETAILED DESCRIPTION:
It is anticipated that 62 participants will be enrolled on to the clinical trial and approximately 100 physicians caring for enrolled participants. There is also a third group that are eligible patients not enrolled in the trial (patients will only be interviewed and will not receive any active treatment) and will not be included in the enrollment numbers or outcome measures.

ELIGIBILITY:
Inclusion Criteria for Clinical trial patients:

1. Patient ≥ 18 to 75 years of age at baseline
2. Diagnosis of ulcerative colitis (verified by a typical clinical history as well as characteristic appearance on endoscopy and histology)
3. Current hospital admission for ulcerative colitis treatment (expecting IV corticosteroid initiation)
4. Meeting the following definition of acute severe ulcerative colitis as defined as having ≥ 4 bowel movements per day with visible blood and one of the following:

   1. Temperature > 37.5C
   2. Pulse > 90 BPM
   3. Hemoglobin < 10.5g/dL
   4. Erythrocyte sedimentation rate ≥ 30mm/h
   5. Weight loss > 5 lbs over 3 months
   6. C-reactive protein ≥ 3.0mg/dL
   7. Fecal calprotectin >782 mg/kg (within 4 weeks)
   8. Oral corticosteroid use for ≥ 14 days at a dose equivalent to ≥ 30mg/day
5. Prior history of receiving at least one dose of adalimumab, certolizumab, infliximab, or golimumab originator or biosimilars
6. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, daily bowel movement symptoms surveys, and other study procedures
7. Evidence of a personally signed and dated informed consent document indicating that the participant (or a legal representative) has been informed of all pertinent aspects of the study
8. Ability to take oral medication and be willing to adhere to the study intervention regimen
9. For females of reproductive potential (i.e., females <55 years of age with intact ovaries and fallopian tubes): A negative pregnancy test on admission and intent to use highly effective contraception during 3-month follow-up period which include the following.

   1. Combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal, injectable) associated with the inhibition of ovulation, initiated at least 30 days prior to study baseline
   2. Progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation, initiated at least 30 days prior to study baseline
   3. Bilateral tubal occlusion/ligation (could be via hysteroscopy, provided a hysterosalpingogram confirmed success of the procedure)
   4. Vasectomized partner(s) provided the vasectomized partner had received medical confirmation of the surgical success and was the sole sexual partner of the trial participant
   5. Intrauterine device or intrauterine hormone-releasing system
   6. Lifestyle abstinence (refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the patient)
   7. Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods)
   8. Consistent use of barrier contraception

Exclusion Criteria for Clinical trial patients:

1. Presence of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, or clinical findings suggestive of Crohn's disease
2. On IV corticosteroids for ≥ 72 hours prior to enrollment continuously (at any institution)
3. Currently pregnant or breastfeeding
4. Patients who meet diagnostic criteria for toxic megacolon during this current admission. This will be determined by the study team and inpatient treatment team according to the following supportive criteria: Having dilation of the colon > 6m and three of the following (Temperature>38C, HR >120 BPM, WBC>10500/µL, Hemoglobin < 10.5mg/dL) and one of the following (dehydration, altered mental status, severe electrolyte disturbances, and hypotension)
5. Known hypersensitivity to any of the following drugs or constituents: methylprednisolone, cyclosporine, tofacitinib, or upadacitinib
6. Patients who had previous exposure to upadacitinib. Previous exposure to other Janus kinase (JAK) inhibitors (eg, tofacitinib, baricitinib, or filgotinib) are permissible.
7. Patients with ongoing severe infection (as determined by the study team), including untreated or inadequately treated latent or active tuberculosis (TB)

   1. Active CMV colitis is defined as having > 5 CMV inclusion bodies per high powered field in any one ulcer at baseline. If CMV colitis is confirmed, the patient can remain in the trial if permissible by the infectious disease and primary treatment team and if concomitant anti-viral therapy is initiated.
   2. Patients with a positive stool exam for enteric pathogens can remain in the trial. Initiation of treatment at the discretion of the treatment team and infectious disease team if needed.
8. Patients who had received any investigational agent or procedure within 30 days or five half-lives prior to baseline, whichever is longer, or were enrolled in an interventional study
9. Current malignancy with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin.
10. Patients who had a history of colectomy (total or subtotal), ileoanal pouch, Kock pouch, or ileostomy or were planning bowel surgery
11. Moderate or severe renal, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, neurological, or psychiatric condition including the following:

    1. Neutropenia - ANC <1200 cells/mm3 or Total white blood cell count <2500/µL
    2. Hemoglobin < 8mg/dL
    3. Platelet count <80,000/µL
    4. Moderate/severe renal impairment with eGFR <30mL/min/1.73m2 (by simplified four-variable Modification of Diet in Renal)
    5. ALT and AST liver biochemistry levels that are ≥ 2 times the upper limit of normal (ULN)
12. Cirrhosis with mild to severe hepatic impairment (defined as a Child-Pugh score ≥5)
13. History of uncontrolled hypertension (systolic blood pressure >160mmHg or diastolic blood pressure > 100mmHg despite anti-hypertensives)
14. Any of the following cardiovascular conditions:

    1. Recent (within previous 6 months) cerebrovascular accident, myocardial infarction, or coronary stenting
    2. Recent (within previous 6 months) moderate-to-severe congestive heart failure (New York Heart Association class III or IV)
15. History of inherited or acquired conditions that predispose to hypercoagulability including the following. Please note, that patients with a remote history of provoked thrombotic event or recent thrombotic event on systemic anticoagulation are NOT exclusionary.

    1. Antiphospholipid syndrome
    2. Factor V Leiden mutation
    3. Prothrombin G20210A mutations
    4. Deficiencies of antithrombin

    f. Deficiency of protein C g. Deficiency of protein S h. Heparin cofactor II deficiency i. Plasminogen and plasminogen activator inhibitor-1 j. Dysfibrinogenemia k. Factor XII deficiency
16. Patients with total cholesterol <80 mg/dL at baseline
17. Patients who had a history of an allergic reaction or significant sensitivity to constituents of the treatment (and its excipients) and/or other products in the same class of medication (ex., tofacitinib)
18. Patients who had hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection defined as:

    1. HBV: hepatitis B surface antigen (HBsAg) positive with detectable deoxyribonucleic acid (DNA) not on therapy. Patients with serologic evidence of a resolved prior HBV infection (i.e., HBsAg-negative and anti-HB Core-positive) or patients with HBsAg positive on suppressive HBV therapy with low DNA (<105 copies/mL or <104 IU/mL negative) are not exclusionary
    2. HCV: HCV ribonucleic acid detectable in any patient with anti-HCV antibody
    3. HIV: Confirmed positive anti-HIV antibody with CD4 counts <350 cells/uL or acquired immunodeficiency syndrome (AIDS)- defining opportunist infection
19. Solid organ or bone marrow transplant within 1 year or expected transplant within 6 months
20. History of more than one episode of herpes zoster, a history of disseminated herpes zoster or disseminated herpes simplex
21. Current use of medications which significantly increase the risk of venous thromboembolic event as determined by the investigator including:

    1. Hormone replacement therapy
    2. Testosterone
    3. Tamoxifen
22. Vaccination with live or attenuated live vaccines within 6 weeks of baseline or scheduled to receive these vaccines during study period or within 140 days (20 weeks) after last dose of study medication.
23. History of any lymphoproliferative disorder (such as EBV-related lymphoproliferative disorder), history of lymphoma, leukemia, myeloproliferative disorders, multiple myeloma, or signs and symptoms suggestive of current hematologic disease.
24. Patients who had a history of spontaneous GI perforation (other than appendicitis or mechanical injury), diverticulitis, or significantly increased risk of GI perforation per investigator's judgement
25. Actively receiving strong CYP3A4 inducers or inhibitors prior to the first dose of study drug or are expected to receive any of these medications during the study period. This includes grapefruit and grapefruit juice.
26. The presence of any condition possibly affecting oral drug absorption (e.g., gastrectomy, clinically significant diabetic gastroenteropathy, or certain types of bariatric surgery such as gastric bypass). Procedures such as gastric banding that simply divide the stomach into separate chambers are NOT exclusionary.
27. Patients who had a history of a clinically significant medical condition or any other reason which, in the opinion of the investigator, would have interfered with the patient's participation in this study, would have made the patient an unsuitable candidate to receive treatment, or would have put the patient at risk by participating in the protocol

Inclusion criteria for Physicians:

1. Clinicians (Internal medicine residents, gastroenterology fellows, and attending gastroenterologists or colorectal surgeons) caring for the patients enrolled in the clinical trial

Exclusion criteria for Physicians:

1. Non-clinicians not caring for the enrolled patient

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of randomly allocated participants to first stage of intervention | Approximately 100 Days (intervention plus 90 days of follow-up)
  The study team will assess the ability of the investigators to execute the SMART, as well as the ability to treat participants with each of three first stages of intervention.
Proportion of randomly assigned patients who completed study period and 90-day follow-up | Up to 100 days (intervention plus follow-up)
  The study team will assess the ability of the investigators to execute the SMART, as well as the ability to treat participants to complete one of the adaptive treatment strategies and complete the SMART study (including the intervention and follow-up period).
Proportion of patients with completed CRP and daily bowel movements recorded on Day 2 or Day 3 prior to sequentially randomized allocation | Day 2 or Day 3 (prior to sequentially randomized allocation)
  To assess the feasibility of using bowel movements and CRP as the study primary tailoring variable to determine if these are too long or burdensome, and if these variables can be obtained in a timely and complete fashion.
Proportion of patients who successfully underwent the second randomization (or transition to the second stage among those not re-randomized) | Up to 10 days
  The study will assess the feasibility of using real-time sequentially randomized allocation performed successfully by the treatment team.
Proportion of patients reporting trial design acceptable | Approximately Day 10 (end of study treatment period)
  This will be measured by semi-structured interviews with patients and clinicians at the end of study period. One question for this outcome will be asked the study was acceptable (yes or no).
Proportion of inpatient physicians reporting trial design acceptable | Approximately Day 10 (end of study treatment period)
  This will be measured by semi-structured interviews with patients and clinicians at the end of study period. One question for this outcome will be asked the study was acceptable (yes or no).
Proportion of patients who complete the trial who successfully underwent the second randomization (non-responders) or continued current therapy (responders) of all enrolled patients. | Up to 100 days (intervention plus follow-up)
  The study team will assess the ability of the investigators to execute the SMART, as well as the ability to treat participants to complete one of the adaptive treatment strategies and complete the SMART study (including the intervention and follow-up period).

SECONDARY OUTCOMES:
Proportion of patients undergoing same-admission colectomy | Approximately 10 days (prior to discharge from index admission)
  Colectomy events prior to discharge from index admission will be recorded as yes/no and compared between adaptive treatment strategies.
Proportion of patients undergoing colectomy within follow-up | Up to 100 days (intervention plus follow-up)
  Colectomy events within follow-up of index admission will be recorded as yes/no and compared between arms.
Incidence and severity of adverse events | Up to 100 days (intervention plus follow-up)
  Incidence and severity of adverse events will be reported. Shingles, acne, major cardiovascular events, venous thromboembolic events, cancers and other infections are adverse events of special interest (AESI). The study team will also record the incidence of serious infections and incidence and severity of laboratory abnormalities between first treatment stage and adaptive treatment strategies.
  Adverse event will be graded as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Proportion of patients in steroid-free remission at 90 days | At 90-day follow-up
  Patients will be assessed for on-going steroid use (any dose) at the 90-day follow-up and will be recorded as yes/no and compared between arms.
Proportion of patients in initial clinical response (C-reactive protein and number of bowel movements) without non-trial rescue therapy or colectomy at 120 hours (5 days) after initiating first stage therapy per to treatment and ATS. | 5 days from randomization
  Patients assessed for initial clinical response, initiation of non-trial rescue therapy, or colectomy with 120 hours from randomization. Initial clinical response is defined by a reduction in bowel movements per 24 hours by ≥ 60% from enrollment or less than 4 bowel movements per day AND a C-reactive protein (CRP) < 1 mg/dL
Proportion of patients without rescue therapy during intervention period or colectomy within 90 days per treatment | Up to 100 days (intervention plus follow-up)
  Patients will be assessed for initiation non-study rescue therapy of at the 90-day follow-up and will be recorded as yes/no and compared between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Berinstein, MD, MSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan includes:
  * de-identified dataset will be placed in a public repository after publication.
Supporting Information: Study Protocol, ICF